CLINICAL TRIAL: NCT04442126
Title: A Phase 1/2 Study of NM21-1480 (Anti-PDL-1/Anti-4-1BB/Anti-HSA Tri-Specific Antibody) in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of NM21-1480 in Adult Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A business decision was made to discontinue further enrollment. There were no safety concerns that contributed to this decision.
Sponsor: Numab Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NB-ND021 (NM21-1480)-101; 2020-0355 (Other: MDACC Protocol ID)
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor; Non-small Cell Lung Cancer; Colorectal Cancer; Squamous Cell Carcinoma; Ovarian Carcinoma; Peritoneal Carcinoma; Fallopian Tube Cancer; Head and Neck Squamous Cell Carcinoma; Triple Negative Breast Cancer
Keywords: Carcinoma; Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Carcinoma, Squamous Cell; Ovarian Neoplasms; Fallopian Tube Neoplasms; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms; Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NM21-1480 Treatment arm (Experimental)
  Interventions: Biological: NM21-1480

INTERVENTIONS:
Biological: NM21-1480 — Trispecific anti-PD-L1/anti-4-1BB/anti-Human Serum Albumin (HSA) single-chain Fv fusion protein

SUMMARY:
This is a first-in-human, open-label, multi-center, Phase 1/2, dose-escalation study with expansion cohorts to evaluate NM21-1480 for safety and immunogenicity, to determine the maximal tolerated dose and recommended Phase 2 dose, define the pharmacokinetics, to explore the pharmacodynamics, and to obtain preliminary evidence of the clinical activity in adult patients with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Patients with any previously treated solid tumor-type other than hepatocellular carcinoma or intrahepatic cholangiocarcinoma that is advanced, or recurrent and progressing since last anti-tumor therapy, and for which no alternative, standard therapy exists.
* Prior chemotherapy, radiation therapy or immunotherapy must have been completed at least 4 weeks prior to the administration of the first dose of study drug, and patient has recovered

Part B:

* Patients with Non-small Cell Lung Cancer (NSCLC) or other protocol specified solid tumors with locally advanced or metastatic, non-resectable disease, which has progressed despite treatment with first-line standard of-care treatment, or first- and second-line treatment, dependent on expansion cohort.
* Prior therapy must have been completed 2-4 weeks prior to the administration of the first dose of study drug as specified per protocol according to type of prior therapy

Exclusion Criteria:

* Patient previously had known immediate or delayed hypersensitivity reaction or idiosyncrasy to the excipients
* Part A: Treatment with any PD-1, or Cytotoxic T-Lymphocyte Associated Protein (CTLA)-4 directed antibody, or with any other immunotherapy within 4 weeks prior to initiation of the study drug.
* Part A: Use of other biological investigational drugs (drugs not marketed for any indication), including use of investigational drugs targeting CD137/4-1BB within at least 5 half-lives (or within 8 weeks, whatever is longer) prior to the administration of the first dose of study drug.
* Part B: As defined per protocol for each expansion cohort, has not been treated with specified first/second-line standard-of-care therapies biological drugs (marketed or investigational) for treatment of the current cancer, or has not adequately recovered from AEs that occurred with prior therapy.
* Patient has an active autoimmune disease or a documented history of autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (14):
  - UCHealth Poudre Valley Hospital, Fort Collins, Colorado
  - Augusta University Medical Center, Augusta, Georgia
  - Tulane University Medical Center, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - Dartmouth Cancer Center, Lebanon, New Hampshire
  - NYU Langone Medical Center - Perlmutter Cancer Center (NYU Cancer Institute), New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - The University Of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Spain (11):
  - Hospital Universitario de A Coruna, A Coruña
  - Hospital Universitario Vall dHebron, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Complejo Hospitalario de Jaen, Jaén
  - Centro Integral Oncologico Clara Campal, Madrid
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Son Llatzer, Palma de Mallorca
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- National Taiwan University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Dose Level 1 NM21-1480-Q2W 0.15mg: Flat dose level; 0.15mg (Dose Level 1)
- Part A Dose Level 2 NM21-1480-Q2W 1.5mg: Flat dose level; 1.5mg (Dose Level 2)
- Part A Dose Level 3 NM21-1480-Q2W 8mg: Flat dose level; 8mg (Dose Level 3)
- Part A Dose Level 4 NM21-1480-Q2W 24mg: Flat dose level; 24mg (Dose Level 4)
- Part A Dose Level 5 NM21-1480-Q2W 80mg: Flat dose level; 80mg (Dose Level 5)
- Part A Dose Level 6 NM21-1480-Q2W 240mg: Flat dose level; 240mg (Dose Level 6)
- Part A Dose Level 7 NM21-1480-Q2W 800mg: Flat dose level; mg800 (Dose Level 7)
- Part A2 NM21-1480-Q2W: This part of the study consisted of a 1400mg flat dose across one cohort.
- Part B NM21-1480-Q2W: This part of the study consisted of a 800mg flat dose across three cohorts.
Period: Overall Study
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Started | 1 | 1 | 3 | 3 | 6 | 3 | 9 | 5 | 21
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 3 | 6 | 3 | 9 | 5 | 21
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 3
Not completed — Death | 1 | 0 | 0 | 1 | 2 | 2 | 4 | 1 | 5
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 10
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Progressive Disease | 0 | 1 | 3 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A Dose Level 1NM21-1480-Q2W0.15mg: Flat dose level; 0.15mg(Dose Level 1)
- Part A Dose Level 2NM21-1480-Q2W1.5mg: Flat dose level; 1.5mg(Dose Level 2)
- Part A Dose Level 3NM21-1480-Q2W 8mg: Flat dose level; 8mg(Dose Level 3)
- Part A Dose Level 4NM21-1480-Q2W24mg: Flat dose level; 24mg(Dose Level 4)
- Part A Dose Level 5NM21-1480-Q2W80mg: Flat dose level; 80mg(Dose Level 5)
- Part A Dose Level 6NM21-1480-Q2W240mg: Flat dose level; 240mg(Dose Level 6)
- Part A Dose Level 7NM21-1480-Q2W800mg: Flat dose level; mg800(Dose Level 7)
- Part A2 NM21-1480-Q2W: This part of the study consisted of a 1400mgflat dose across one cohort.
- Part B NM21-1480-Q2W: This part of the study consisted of a 800mgflat dose across three cohorts.
- Total: Total of all reporting groups
Arm/Group | Part A Dose Level 1NM21-1480-Q2W0.15mg | Part A Dose Level 2NM21-1480-Q2W1.5mg | Part A Dose Level 3NM21-1480-Q2W 8mg | Part A Dose Level 4NM21-1480-Q2W24mg | Part A Dose Level 5NM21-1480-Q2W80mg | Part A Dose Level 6NM21-1480-Q2W240mg | Part A Dose Level 7NM21-1480-Q2W800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 3 | 9 | 5 | 21 | 52
Age, Categorical [Count of Participants; unit: Participants] — Count of Participants Unit of Measure: Participants
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 1 | 0 | 2 | 2 | 3 | 2 | 7 | 3 | 9 | 29
    >=65 years | 0 | 1 | 1 | 1 | 3 | 1 | 2 | 2 | 12 | 23
Sex: Female, Male [Count of Participants; unit: Participants] — Count of Participants Unit of Measure: Participants
  Participants
    Female | 0 | 1 | 2 | 2 | 2 | 1 | 3 | 1 | 8 | 20
    Male | 1 | 0 | 1 | 1 | 4 | 2 | 6 | 4 | 13 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Count of Participants Unit of Measure: Participants
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Not Hispanic or Latino | 1 | 1 | 3 | 3 | 6 | 3 | 9 | 5 | 20 | 51
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Count of Participants Unit of Measure: Participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 4
    White | 0 | 0 | 3 | 2 | 5 | 3 | 6 | 5 | 20 | 44
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v5.0
Description: Frequency and severity of adverse events
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Participant with any TREA
Measure: Number; unit: participants
Groups:
- Part A Dose Level 1 NM21-1490-Q2W 0.15mg: Part A Dose Level 1 NM21-1490-Q2W 0.15mg
- Part A Dose Level 2 NM21-1490-Q2W 1.5mg: Part A Dose Level 2 NM21-1490-Q2W 1.5mg
- Part A Dose Level 3 NM21-1490-Q2W 8mg: Part A Dose Level 3 NM21-1490-Q2W 8mg
- Part A Dose Level 4 NM21-1490-Q2W 24mg: Part A Dose Level 4 NM21-1490-Q2W 24mg
- Part A Dose Level 5 NM21-1490-Q2W 80mg: Part A Dose Level 5 NM21-1490-Q2W 80mg
- Part A Dose Level 6 NM21-1490-Q2W 240mg: Part A Dose Level 6 NM21-1490-Q2W 240mg
- Part A Dose Level 7 NM21-1490-Q2W 800mg: Part A Dose Level 7 NM21-1490-Q2W 800mg
- Part A2 NM32-1480-Q2W: Part A2 NM32-1480-Q2W 1400mg
- Part B NM32-1480-Q2W: Part B NM32-1480-Q2W 800mg
Arm/Group | Part A Dose Level 1 NM21-1490-Q2W 0.15mg | Part A Dose Level 2 NM21-1490-Q2W 1.5mg | Part A Dose Level 3 NM21-1490-Q2W 8mg | Part A Dose Level 4 NM21-1490-Q2W 24mg | Part A Dose Level 5 NM21-1490-Q2W 80mg | Part A Dose Level 6 NM21-1490-Q2W 240mg | Part A Dose Level 7 NM21-1490-Q2W 800mg | Part A2 NM32-1480-Q2W | Part B NM32-1480-Q2W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 3 | 9 | 5 | 21
participants | 1 | 1 | 3 | 3 | 5 | 3 | 9 | 5 | 16

2. Primary Outcome: Maximum Tolerated Dose (MTD) of NM21-1480
Description: To determine the MTD of NM21-1480 based on Part A. Note, No MTD was identified across all dose levels tested and a technical MTD was defined by the SMC as 800 mg following Part A, which was updated to 1400 mg by the SMC after completion of Part A-2.
Time Frame: Cycle 1 (28 days).
Population: MTD of NM21-1480 based on Part A and part A2. No MTD was identified across all dose levels tested and a technical MTD was defined by the SMC as 800 mg following Part A, which was updated to 1400 mg by the SMC after completion of Part A-2.
Measure: Number; unit: mg
Groups:
- Part A Dose Level 1 NM21-1480-Q2W 0.15mg: Part A Dose Level 1 NM21-1480-Q2W 0.15mg
- Part A Dose Level 2 NM21-1480-Q2W 1.5mg: Part A Dose Level 2 NM21-1480-Q2W 1.5mg
- Part A Dose Level 3 NM21-1480-Q2W 8mg: Part A Dose Level 3 NM21-1480-Q2W 8mg
- Part A Dose Level 4 NM21-1480-Q2W 24mg: Part A Dose Level 4 NM21-1480-Q2W 24mg
- Part A Dose Level 5 NM21-1480-Q2W 80mg: Part A Dose Level 5 NM21-1480-Q2W 80mg
- Part A Dose Level 6 NM21-1480-Q2W 240mg: Part A Dose Level 6 NM21-1480-Q2W 240mg
- Part A Dose Level 7 NM21-1480-Q2W 800mg: Part A Dose Level 7 NM21-1480-Q2W 800mg
- Part A2 NM21-1480-Q2W 1400mg: Part A2 NM21-1480-Q2W 1400mg
- Part B NM21-1480-Q2W 800mg: Part B NM21-1480-Q2W 800mg
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W 1400mg | Part B NM21-1480-Q2W 800mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 5 | 0
mg |  |  |  |  |  |  | 800 | 1400 |

3. Primary Outcome: Determination of Phase 2 Dose of NM21-1480
Description: To determine the recommended Phase 2 dose of NM21-1480 for Part B of the study
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Measure: Number; unit: mg
Arm/Group | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W 1400mg
Number analyzed (Participants) | 26 | 5
mg | 800 | 800

4. Primary Outcome: To Determine the Anti-tumor Activity (Best Overall Response) of NM21-1480 According to RECIST 1.1
Description: For best overall response (BOR) and objective response rate (ORR), patients in the Efficacy Analysis Set (EAS) who did not have sufficient on-study tumor assessments to characterize response were included in the denominator when calculating BOR percent and ORR and were thus treated as non-responders.
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: The ORR for each given group (dose level, cohort, or arm) in the EAS are summarized according to RECIST 1.1 (and according to iRECIST), accompanied by a 2-sided exact 95% Clopper-Pearson confidence interval (CI).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W 1400mg | Part B NM21-1480-Q2W 800mg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 3 | 9 | 5 | 21
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Assessment of the Maximum Observed Serum Concentration Determined by Direct Inspection of the Concentration Versus Time Data (Cmax)
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Cmax determined at C1 for all dose levels with the exception of Part A Dose Level 1 which has been noted as NA ,for which was BLQ. Lower limit of quantification (LLOQ) of NM21-1480 = 5 ng/mL.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 3 | 8 | 4 | 9
ng/mL | NA (NA) — BLQ | 184.3 (184.3) | 1604 (1101) | 6334 (2331) | 19800 (5576) | 66890 (43340) | 204700 (32070) | 420300 (12040) | 258500 (65390)

6. Secondary Outcome: Assessment of the the Minimum Observed Serum Concentration Determined by Direct Inspection of the Concentration Versus Time Data (Cmin)
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Cmin determined at C1 for all dose levels with the exception of Part A Dose Level 1 which has been noted as NA ,for which was BLQ. Note: Lower limit of quantification (LLOQ) of NM21-1480 = 5 ng/mL.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 3 | 8 | 4 | 9
ng/mL | NA (NA) — BLQ | 0 (0) | 201.7 (227.5) | 658.2 (451.7) | 4203 (1340) | 15880 (14540) | 48670 (17090) | 166000 (41730) | 54270 (22000)

7. Secondary Outcome: Assessment of the Time From Dosing at Which Cmax is Apparent Determined by Direct Inspection of the Concentration Versus Time Data (Tmax)
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Tmax determined at C1 for all dose levels with the exception of Part A Dose Level 1 and Part A Dose Level 2. Lower limit of quantification (LLOQ) of NM21-1480 = 5 ng/mL.
Measure: Mean (Full Range); unit: h
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 3 | 8 | 4 | 9
h | NA [lower limit NA] — BLQ | 1 [1 to 1] | 26.533 [1 to 77.58] | 6.407 [4.92 to 8.03] | 5.778 [0.97 to 25.37] | 2.340 [0.95 to 5.05] | 8.720 [1.50 to 48.60] | 3.13 [1.53 to 8.58] | 1.587 [1.53 to 1.7]

8. Secondary Outcome: Assessment of the Terminal Phase (Apparent Elimination) Rate Constant (λz)
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Lambda z determined at C1 for all dose levels with the exception of Part A Dose Level 1,2 and 3. Lower limit of quantification (LLOQ) of NM21-1480 = 5 ng/mL. The constant Lambda z and its derived parameters meet one of the following conditions: the adjusted regression coefficient is less than 0.8 or the AUC%extrap exceeds 20%.
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 5 | 3 | 8 | 4 | 4
1/h |  |  |  | 0.007163 (0.002300) | 0.005417 (0.002940) | 0.003352 (0.001460) | 0.003522 (0.0007292) | 0.002923 (0.001239) | 0.002840 (0.0006234)

9. Secondary Outcome: Assessment of the Elimination Half-life (t½)
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Assessment of the elimination half-life (t½) determined at C1 for all dose levels with the exception of Part A Dose Level 1, Part A Dose Level 2 and Part A Dose Level 3. Lower limit of quantification (LLOQ) of NM21-1480 = 5 ng/mL. No descriptive statistics determined when fewer than three individual PK parameters are available.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 5 | 3 | 8 | 4 | 4
h |  |  |  | 102.824 (28.4100) | 165.179 (90.7037) | 230.048 (80.2781) | 203.241 (36.4457) | 272.095 (116.9242) | 253.230 (56.1072)

10. Secondary Outcome: Assessment of the Area Under the Serum Concentration-time Curve Extrapolated From the Last Quantifiable Concentration to Infinity Quantifiable Concentration to Infinity (AUC[0-infinity])
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: AUC0-t determined at C1 for all dose levels with the exception of Part A Dose Level 1 and Part A Dose Level 2. Lower limit of quantification (LLOQ) of NM21-1480 = 5 ng/mL.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 0 | 0 | 3 | 3 | 6 | 3 | 8 | 4 | 9
h*ng/mL |  |  | 81570 (59740) | 802200 (339000) | 2602000 (1177000) | 9442000 (6364000) | 32630000 (3717000) | 57570000 (12480000) | 39560000 (12150000)

11. Secondary Outcome: Assessment of the Area Under Serum Concentration-time Curve Over Dosing Interval (AUCtau)
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: AUCtau determined at C1 for all dose levels with the exception of Part A Dose Level 1, Part A Dose Level 2 and Part A Dose Level 3. Lower limit of quantification (LLOQ) of NM21-1480 = 5 ng/mL.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 6 | 3 | 8 | 4 | 7
h*ng/mL |  |  |  | 803200 (340000) | 2662000 (1022000) | 9648000 (6863000) | 32420000 (3342000) | 69890000 (3413000) | 36810000 (11890000)

12. Secondary Outcome: Assessment of the Clearance (CL)
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Assessment of the clearance (CL) determined at C1 for all dose levels with the exception of Part A Dose Levels 1, 2 and 3. Lower limit of quantification (LLOQ) of NM21-1480 = 5 ng/mL.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 5 | 3 | 8 | 4 | 4
L/h |  |  |  | 0.03037 (0.01332) | 0.03034 (0.01764) | 0.02257 (0.01329) | 0.01717 (0.002606) | 0.01218 (0.002768) | 0.01596 (0.004527)

13. Secondary Outcome: Assessment of the Volume of Distribution (Vd)
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Assessment of the volume of distribution (Vd) determined at C1 for all dose levels with the exception of Part A Dose Level 1,2 and 3. Lower limit of quantification (LLOQ) of NM21-1480 = 5 ng/mL.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 5 | 3 | 8 | 4 | 4
L |  |  |  | 4.155 (0.9071) | 5.882 (2.263) | 6.674 (3.379) | 4.952 (0.6848) | 4.454 (0.9507) | 5.930 (2.472)

14. Secondary Outcome: Assessment of the Frequency of Specific Anti-drug Antibodies to NM21-1480
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: A patient is considered positive if they are positive at any scheduled or unscheduled post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W 1400mg | Part B NM21-1480-Q2W 800mg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 3 | 9 | 5 | 21
Participants | 1 | 1 | 2 | 3 | 5 | 3 | 6 | 1 | 14

15. Secondary Outcome: To Determine the Anti-tumor Activity (Duration of Response) of NM21-1480 According to RECIST 1.1
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Where blank the duration of response was not evaluable.
Measure: Median (Full Range); unit: Months
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Months |  |  |  | 1.84 [1.84 to 1.84] |  |  |  |  |

16. Secondary Outcome: To Determine the Anti-tumor Activity (Time-to-response) of NM21-1480 According to RECIST 1.1
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: One patient at dose level 4 exhibited a PR (Partial Response).
Measure: Number; unit: Days
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Days |  |  |  | 110 |  |  |  |  |

17. Secondary Outcome: To Determine the Anti-tumor Activity (Progression-free Survival) of NM21-1480 According to RECIST 1.1
Time Frame: From baseline to up to 12 weeks post last dose, up to 48 weeks.
Population: Progression-Free Survival (PFS) is defined as the time from the start of study treatment until the earliest documented date of disease progression or death.
  [1] Q1, Median and Q3 are Kaplan-Meier estimates and the 2-sided 95% confidence interval for median is calculated using the Brookmeyer-Crowley method.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
Number analyzed (Participants) | 0 | 0 | 3 | 3 | 5 | 2 | 7 | 0 | 19
Months |  |  | 1.84 [1.708 to 3.253] | 5.49 [5.454 to 5.552] | 1.81 [0.657 to 9.002] | 7.28 [3.548 to 11.006] | 2.86 [1.314 to 7.261] |  | 1.41 [0.0526 to 2.727]

ADVERSE EVENTS:
Time Frame: Up to 3 years.
Description: The safety population included all participants enrolled in the study who received at least one dose of study treatment.
Arm/Group | Part A Dose Level 1 NM21-1480-Q2W 0.15mg | Part A Dose Level 2 NM21-1480-Q2W 1.5mg | Part A Dose Level 3 NM21-1480-Q2W 8mg | Part A Dose Level 4 NM21-1480-Q2W 24mg | Part A Dose Level 5 NM21-1480-Q2W 80mg | Part A Dose Level 6 NM21-1480-Q2W 240mg | Part A Dose Level 7 NM21-1480-Q2W 800mg | Part A2 NM21-1480-Q2W | Part B NM21-1480-Q2W
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 0/3 | 0/6 | 0/3 | 0/9 | 0/5 | 1/21
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 1/3 | 1/3 | 2/6 | 1/3 | 4/9 | 3/5 | 6/21
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 3/3 | 5/6 | 3/3 | 9/9 | 5/5 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Dose Level 1 NM21-1480-Q2W 0.15mg (N=1) | Part A Dose Level 2 NM21-1480-Q2W 1.5mg (N=1) | Part A Dose Level 3 NM21-1480-Q2W 8mg (N=3) | Part A Dose Level 4 NM21-1480-Q2W 24mg (N=3) | Part A Dose Level 5 NM21-1480-Q2W 80mg (N=6) | Part A Dose Level 6 NM21-1480-Q2W 240mg (N=3) | Part A Dose Level 7 NM21-1480-Q2W 800mg (N=9) | Part A2 NM21-1480-Q2W (N=5) | Part B NM21-1480-Q2W (N=21)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Dose Level 1 NM21-1480-Q2W 0.15mg (N=1) | Part A Dose Level 2 NM21-1480-Q2W 1.5mg (N=1) | Part A Dose Level 3 NM21-1480-Q2W 8mg (N=3) | Part A Dose Level 4 NM21-1480-Q2W 24mg (N=3) | Part A Dose Level 5 NM21-1480-Q2W 80mg (N=6) | Part A Dose Level 6 NM21-1480-Q2W 240mg (N=3) | Part A Dose Level 7 NM21-1480-Q2W 800mg (N=9) | Part A2 NM21-1480-Q2W (N=5) | Part B NM21-1480-Q2W (N=21)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 4 (4) — General disorders and administration site conditions
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) — General disorders and administration site conditions
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) — General disorders and administration site conditions
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — General disorders and administration site conditions
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General disorders and administration site conditions
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight fluctuation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroxine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmondry embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chlongitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stoma site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Hyperthyroidism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinal odema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT04442126/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04442126/SAP_001.pdf